CLINICAL TRIAL: NCT03523325
Title: Recovery of Symptoms, Function, Tendon Structure and Mechanical Properties in Patients With Achilles Tendinopathy: A Comparison Between Men and Women
Brief Title: Achilles Tendinopathy, Treatment With eXercise Comparing Men and Women
Acronym: ATX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AR072034-01A1 (NIH)
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Achilles Tendinopathy; Achilles Tendonitis; Achilles Tendon Pain; Achilles Degeneration; Achillodynia
Keywords: Tendinopathy; Tendon; Rehabilitation; Exercise treatment
MeSH Terms: conditions — Tendinopathy | interventions — Exercise Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: One intervention with comparison between males and females
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise treatment — Treatment protocol is an exercise program consisting of four different phases (Silbernagel protocol). The progression consists of increasing number of repetitions, resistance, speed and range of motion of the exercises. A pain-monitoring model is used to adjust the exercise loads and progression through the four phases.
  Other Names: Rehabilitation exercise; Physical Therapy treatment

SUMMARY:
This study will evaluate if there is a difference in recovery of tendon structure and mechanical properties between males and females with Achilles tendinopathy receiving exercise treatment. It will evaluate recovery of tendinopathy with exercise intervention using outcome measures for tendon structure and mechanical properties along with validated measures of muscle-tendon function and symptoms.

DETAILED DESCRIPTION:
Achilles tendinopathy has an incidence rate of 2.35 per 1000 in the general population and is most prevalent in middle-aged individuals (35-55 y/o), but occurs in men and women of all ages. The primary symptom is pain during daily activities such as walking and exercising such as running. Aside from the pain, Achilles tendinopathy has been shown to significantly decrease physical activity level, resulting in further negative effects on overall health and well-being. The treatment for Achilles tendinopathy with the highest level of evidence is eccentric exercise, providing mechanical loading of the muscle-tendon unit. In a recent systematic review, all studies reported significant improvements in patient-reported symptoms but at 12 weeks the means ranged from 69-80 (100 being fully recovered) indicating that even with the most effective treatment individuals continued to have symptoms. At this time, other more invasive interventions such as injection therapies (ex. platelet-rich plasma) and surgery are recommended for patients who fail exercise treatment despite a lack of understanding of what factors are related to continued problems. Just achieving a reduction in pain and symptoms with treatment also does not ensure resolution of the tendon's structural abnormalities. In fact, studies evaluating the recovery of tendon structure with exercise suggest that at least 24 weeks may be needed to observe a significant change. Other individual factors such as sex, degree of tendon structural damage and functional deficits are also proposed to influence both the time course and success rate of recovery. The long-term goal of our research is to advance understanding of tendon injuries and repair, enabling tailored treatments to be developed. This study begins to address this long-term goal by evaluating the time-course of recovery in terms of tendon structure (ultrasound imaging) and viscoelastic properties (elastography) along with symptoms (patient-reported outcomes) and muscle-tendon function (functional test-battery) in males and females with Achilles tendinopathy treated with an exercise program. Aim 1 is to evaluate if there are differences in change over time in symptoms, muscle-tendon function, tendon structure, and mechanical properties between males and females with Achilles tendinopathy receiving exercise treatment. Aim 2 is to investigate whether the presence and magnitude of tendon structural abnormality at baseline will affect the ability and time-course of recovery with exercise treatment for Achilles tendinopathy. Aim 3 is to explore if patients who continue to have symptoms at the 16-week evaluation will further improve in symptoms, muscle-tendon function, tendon structure and mechanical properties over the course of one year.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of midportion Achilles tendinopathy

Exclusion Criteria:

* Previous Achilles tendon rupture
* Diagnosis of only insertional Achilles tendinopathy or bursitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Symptoms | Change over time during 12 months with evaluation every 8 weeks
  Victorian Institute of Sports Assessment - Achilles questionnaire (VISA-A), Scale 0-100 with higher scores indicate better outcome.
Tendon Structure | Change over time during 12 months with evaluation every 8 weeks
  Ultrasound imaging of tendon structure
Tendon Mechanical Properties | Change over time during 12 months with evaluation every 8 weeks
  Use of Continuous shear wave elastography to measure shear modulus and viscosity
Muscle-tendon function | Change over time during 12 months with evaluation every 8 weeks
  Functional test battery consisting of one endurance heel-rise test and three jump tests

SECONDARY OUTCOMES:
Activity level | Change over time during 12 months with evaluation every 8 weeks
  Measure of daily step counts
Foot and Ankle related quality of life | Change over time during 12 months with evaluation every 8 weeks
  Foot and Ankle Outcome Score (FAOS) Quality of Life subscale, scale ranges from 0-100 with higher score indicate better outcome.
Kinesiophobia | Change over time during 12 months with evaluation every 8 weeks
  Tampa Scale of Kinesiophobia (TSK), scale ranges from 17 to 68 where the higher scores indicate an increasing degree of kinesiophobia.
Physical Activity level | Change over time during 12 months with evaluation every 8 weeks
  Physical Activity Scale (PAS), scale ranges from 1-6 with higher score indicting greater degree of physical activity.
Pain level | Change over time during 12 months with evaluation every 8 weeks
  Numeric Pain rating scale, scale ranges from 0-10 with higher scores indicating greater degree of pain.
General Health Status- Health related Quality of Life | Change over time during 12 months with evaluation every 8 weeks
  Patient-Reported Outcomes Measurement Information System® (PROMIS) - 29, measures health-related quality of life consisting of 29 question survey divided into seven sub-domains of function including physical functioning, social function, pain interference, pain intensity, sleep, depression, and anxiety.
Mechanical Pain Threshold | Change over time during 12 months with evaluation every 8 weeks
  Pressure Pain Threshold

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smitheman HP, Lundberg M, Harnesand M, Gelfgren S, Gravare Silbernagel K. Putting the fear-avoidance model into practice - what can patients with chronic low back pain learn from patients with Achilles tendinopathy and vice versa? Braz J Phys Ther. 2023 Sep-Oct;27(5):100557. doi: 10.1016/j.bjpt.2023.100557. Epub 2023 Nov 4. PMID 37952338
- [Derived] Hanlon SL, Pohlig RT, Silbernagel KG. Differences in Recovery of Tendon Health Explained by Midportion Achilles Tendinopathy Subgroups: A 6-Month Follow-up. J Orthop Sports Phys Ther. 2023 Apr;53(4):217-234. doi: 10.2519/jospt.2023.11330. Epub 2023 Jan 23. PMID 36688719
- [Derived] Sigurethsson HB, Couppe C, Silbernagel KG. Data driven model of midportion achilles tendinopathy health created with factor analysis. BMC Musculoskelet Disord. 2022 Aug 3;23(1):744. doi: 10.1186/s12891-022-05702-1. PMID 35922770